CLINICAL TRIAL: NCT06064994
Title: The Impact Of Mindfulness Meditation On Pain, Quality Of Sleep, Self-Esteem In Patients With End-Stage Renal Disease Undergoing Hemodialysis In Jordan
Brief Title: Impact Of Mindfulness Meditation On Pain, Quality Of Sleep, Self-Esteem
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hossam Najjem Alhawatmeh, Associate professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 48-2023
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: ESRD
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: An experimental randomized repeated-measures, parallel control design
Who Masked: Outcomes Assessor
Masking Description: A research assistant, who was not involved in any other aspects of the study and was blinded to the randomized allocation, measured the study variables at three points of time
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Patients with ESRD receiving mindfulness meditation
  Interventions: Behavioral: Mindfulness meditation
- Control group (No Intervention): Patients with ESRD receiving traditional care.

INTERVENTIONS:
Behavioral: Mindfulness meditation — The experimental group received the Smith's version of the mindfulness meditation (Smith, 2005), which is a standardized theory-based intervention found to be effective in improving the different dimensions of health. The Smith's version of the mindfulness meditation (Smith, 2005), includes the following components:
  1. Being mindful of breathing (5 minutes).
  2. Being mindful of the body (5 minutes).
  3. Being mindful of thought (5 minutes).
  4. Being mindful of sounds (5 minutes).
  5. Being mindful of taste (5 minutes)
  6. Full meditation
  Other Names: Mindfulness-based intervention
  Arms: Experimental Group

SUMMARY:
Background: Hemodialysis affects patients' lives and is associated with social, occupational, psychological, and societal problems. Mind-body interventions (MBIs), like mindfulness meditation, have been gaining popularity in the health sector. Pain, sleep quality, and self-esteem have all been positively impacted by MBIs in patients with end-stage renal disease (ESRD). Health care providers may be able to provide more thorough care if they are aware of these interventions.

Purpose: To assess the impact of mindfulness meditation on pain, quality of sleep, and self-esteem, and self-management in patients with ESRD undergoing hemodialysis in Jordan.

Methods: An experimental repeated measure, randomized, parallel control design was conducted on 60 patients with ESRD undergoing hemodialysis between March and June 2023 in the dialysis center at Alkarak governmental hospital, Jordan. Participants were randomly assigned to the experimental (N =30) and control groups (N =30) using a simple random assignment method. The experimental group practiced mindfulness meditation for 30 minutes three times per week for five weeks during their hemodialysis treatments. The control group's patients continued to receive hemodialysis treatment as usual, with three hemodialysis sessions for five weeks without any additional intervention. The study variables for both groups were measured at baseline (T0), two weeks after intervention (T1), and at the end of intervention (T2). Variables were measured by the Numeric Pain Rating Scale (NPRS), the Pittsburgh Sleep Quality Index (PSQI), and the Rosenberg Self-Esteem Scale (RSES-M) questionnaire. Descriptive statistics like frequency, mean, and standard deviation were used to describe participants. The repeated measures ANOVA (within-subject) tests were used to examine the study hypotheses.

DETAILED DESCRIPTION:
Problem Statement

Despite the improvements in nursing management and the creation of new facilities, the gold standard treatments for patients with ESRD have not been firmly established (Wen et al., 2021). A significant number of stressors that hemodialysis patients suffer go unsolved during their dialysis treatments (Shinde & Mane, 2014). These stressors, both physical and mental, have a negative impact on physical and psychological health (Jeong & Park, 2012). For this population, how to cope with stressors matters because it can lead to increased morbidity or even earlier death.

Pain and poor sleep quality are highly prevalent among ESRD patients receiving hemodialysis. It has been found that approximately 94.6% and 89.23% of them had poor sleep quality and pain, respectively (Darvishi et al., 2019). Poor Sleep quality and pain among these patients impair not only quality of life, but also immune function. Further, they are even considered risk factors for many other chronic illnesses, significantly increasing morbidity and mortality (Alradaydeh & Khalil, 2019) . Low self-esteem is a major problem in ESRD patients receiving hemodialysis. Low self-esteem has been found to decreases adherence to treatment and self-care behaviors, worsening sleep quality and pain among these patients (Poorgholami et al., 2016).

Mind-body interventions have been employed in other chronic disorders like cancer, irritable bowel syndrome, and coronary heart disease much more than in renal disease (Bennett et al., 2017). Recently, studies that address mind-body interventions, such as relaxation therapy, might exist, but there have been limited studies to investigate the impact of mindfulness meditation. For example, there were studies addressing the effects of the Benson relaxation technique on pain and quality of life in patients on hemodialysis (Rambod et al., 2014). So, those researchers recommended that more research is needed to identify the impacts of mindfulness meditation on pain, quality of sleep, and self-esteem. So, the purpose of this study is to assess the impacts of mindfulness meditation on the mentioned variables among patients undergoing hemodialysis in Jordan.

Significance of the study

There is evidence that enhancing stress coping leads to higher emotional, social, and psychological well-being. However, research on mind-body techniques like mindfulness has attracted both clinical and academic interest (Al-ghabeesh et al., 2021). Mindfulness is seen in Jordan as a socially and culturally acceptable psychotherapy that enhances the psychological well-being of various therapeutic populations (Rayan & Ahmad, 2018). Noteworthy, there are few studies on the effectiveness of mindfulness meditation on sleep quality, pain and self-esteem (Rambod et al., 2014) for patients receiving hemodialysis. Thus, the current study aimed to investigate the impact of mindfulness meditation on pain, quality of sleep, and self-esteem.

The goal of mindfulness meditation is to make it easier for people to cope with the stressors associated with having a chronic condition, such as ESRD. Notably, the growing evidence supporting the use of mindfulness meditations to improve psychological and physical health problems in various healthy and ill populations (Bennett et al., 2017). In ESRD patients undergoing hemodialysis, several studies were conducted to examine the effects of mindfulness meditation on different psychological health problems facing patients undergoing hemodialysis, such as stress, emotion regulation, depression, anxiety, and quality of life ( Alhawatmeh et al., 2021; Pai et al., 2009; Fathi et al., 2020; Dehghan et al., 2020). Theoretically, there were limited studies designed to assess the impact of mindfulness meditation on physical symptoms such as pain and quality of sleep among patients receiving hemodialysis.

Despite the positive effects of meditation on ESRD, further research studies utilizing attempted mindfulness meditation protocol are required. This study aims to investigate the effect of mindfulness-based interventions in patients with ESRD on hemodialysis and to identify the methodological quality of the current literature to support future studies in order to advance knowledge on the topic (Razzera et al., 2021). Hence, results from this study will support a body of knowledge, improve complementary health care, and enhance policy makers in different health settings to employ MBIs modalities such as mindfulness meditation, which improve disease satisfaction.

Purpose of the Study

The purpose of this study is to assess the impact of mindfulness meditation on pain, quality of sleep, and self-esteem in ESRD patients undergoing hemodialysis in Jordan.

Methods

Study Design

An experimental randomized repeated-measures, parallel control design was conducted between April and June 2023 in the dialysis center at Alkarak governmental hospital, Jordan.

Setting

There were 81 working dialysis units distributed all over Jordan. 37 units (46%) administered by the Ministry of Health (MOH), 12 units (15%) administered by Royal Medical Services (RMS), and 2 units (2%) administered by university hospitals. The total number of dialysis machines (944) in all units was distributed as follows: 441 (47%) machines in MOH units, 86 (9%) machines in RMS, 32 (3%) machines in university hospitals, and 385 (41%) machines in private sector hospitals. The overall prevalence per million population in Jordan is 974.86/1,000,000; the highest percent was found in Amman governorate (42.5%); according to the North region, Alkarah has the highest percent with (4.5%), divided into three dialysis units: King Ali Hospital (RMS), Alkarak Government Hospital (MOH), and Italian Hospital (private sector). Alkarak Governmental Hospital, which followed the Ministry of Health and was the primary dialysis unit in South Jordan, served as the data collection site. The unit has 17 machines, has an isolation ward and a regular ward (no isolation), and manages on average between 30 and 35 patients per day.

3.3 Sample

The target population is all patients diagnosed with end-stage renal disease (ESRD) and undergoing hemodialysis in Jordan. The accessible population is the ESRD patients receiving hemodialysis in the Alkarak government hospital (Jordan). A sufficient sample size consisted of 58 participants, selected using a convenience, non-probability sampling method. The G*Power (3.1 software's) analysis suggested that a sample size of 36 participants would be adequate based on a mixed-design (within groups and between groups) repeated measures ANOVA, a power level of 0.95, a significant alpha level of.05, and a moderate effect size of 0.25. A 60% attrition rate was expected in a mostly similar study (Alhawatmeh et al., 2022; Nassim et al., 2021). With a 60% attrition rate anticipated, approximately 24 additional subjects should be included, making up the final sample size of 60 participants.

The inclusion criteria required in this study were being an ESRD patient receiving hemodialysis three times per week, being at least 18 years old, and being able to read and write Arabic. Patients with cognitive dysfunction or mental retardation or those who regularly used psychopharmacological, pain or sleeping pills or received psychotherapy were excluded.

3.4 Study Instruments The data collection tool in this study was a self-reported questionnaire, which consisted of four parts. Part 1 was the demographic data sheet, and Part 2 was the Arabic version of the Numerical Pain Rating Scale (NPRS); and Part 3 was the Arabic version of the Pittsburgh Sleep Quality Index (PSQI).

3.4.1 Demographic Data Sheet

This part included questions for each of the following variables: age, gender, marital status, length of ESRD suffering, smoking status, educational attainment, employment situation, income level, and any comorbidities.

3.4.2 The Numerical Rating Scale (NPRS)

The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain severity in adults (Child et al.,2005).The NPRS is a segmented numerical version of the visual analog scale (VAS), in which the respondent chooses a number (0-10 integers) that best describes the degree of pain (Rodriguez, 2001). Both literate and illiterate rheumatoid arthritis patients have shown high test-retest reliability (r = 0.96 and 0.95, respectively). In patients with chronic pain disorders (pain lasting more than six months), the NPRS was found to have a strong association with the VAS for construct validity, with correlations ranging from 0.86 to 0.95 (Ferraz et al.,1990). For evaluating pain levels in Arabic countries, the Arabic Numeric Pain Rating Scale was a valid and reliable tool.The Arabic Numerical Pain Rating Scale had a high correlation coefficient (r140.93-0.94) with the VAS and VRS.indicating strong consistency in pain level measures among the three pain scales (Alghadir, Anwer, & Iqbal, 2016).

3.4.3 The Pittsburgh Sleep Quality Index (PSQI)

A self-rating questionnaire called the PSQI was created in 1989 by Buysse, Reynolds, Monk, Berman, and Kupfer. The PSQI was created to assess the clinical population's sleep quality. Subjective sleep quality (1 item), sleep latency (2 items), sleep duration (1 item), habitual sleep efficiency (3 items), sleep disturbances (9 items), use of sleeping medication (1 item), and daytime dysfunction (2) are the seven dimensions of sleep characteristics included in the PSQI. The scoring of PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21) Higher score indicate worse sleep quality (Buysse et al., 1989). Internal consistency (Crobach's alpha = 0.85), test-retest reliability (r = 0.85; p value of 0.001), sensitivity of 89.6%, and specificity of 8.65 were all demonstrated by the original English version of the PSQI scale (Buysse et al., 1989). The Arabic PSQI's Cronbach's alpha coefficient was 0.77, indicating acceptable reliability. For evaluating patients who speak Arabic's sleep quality, the Arabic version of the PSQI showed adequate reliability and validity(Alghadir et al., 2016).

3.4.4 Rosenberg Self-Esteem Scale (RSES-M)

The Rosenberg self-esteem scale most frequently used in social science research is the Rosenberg Self-Esteem Scale. Self-esteem is a general assessment of one's value or worth, whether it is good or negative (Rosenberg, 1989). Scoring can be a little challenging because the RSE is a Guttman scale. Responses from people with low self-esteem are "strongly disagree" or "disagree" on things 1, 3, 4, 7, and 10, and "agree" or "strongly agree" on items 2, 5, 6, and 8. Items 3, 7, and 9 are scored as one item if two or three of the three correct answers are provided. Items 1, 8, and 10 are scored as individual items, and combined correct responses (one or two out of two) to items 2 and 6 are considered single things. One or two out of the two correct answers for items 4 and 5 are considered single items. After reversing the scores for the items with negative wording, the scale can alternatively be scored by adding up each 4-point item individually. Total score range from 10-40, highest score reveals better self-esteem (Rosenberg, 1979).

The RSE exhibits excellent internal consistency with a coefficient of repeatability of.92. Over a period of two weeks, test-retest reliability shows correlations of.85 and.88, showing outstanding stability. Validity: uses well-known groups to demonstrate contemporaneous, predictive, and construct validity. The Coopersmith Self-Esteem Inventory and the RSE exhibit strong correlations with one another (Rosenberg, 1979). The Arabic version of the RSES is valid, reliable, and beneficial to use among the Arab community, according to two studies conducted among the Arab population in Jordan and Lebanon (Bezri et al., 2022).

3.5 Intervention

The experimental group received the Smith's version of the mindfulness meditation (Smith, 2005), which is a standardized theory-based intervention found to be effective in improving the different dimensions of health. The Smith's version of the mindfulness meditation (Smith, 2005), includes the following components:

1. Being mindful of breathing: Easily taking in a full, deep breath, filling lungs and simply exhaling, and then breathing naturally. Noticing and simply attending to the air, as it flows in and out of nose and moves deeper into throat and lung (5 minutes).
2. Being mindful of the body: Attending to how the body feels from head to toes, and noticing whatever sensations come and go. Whenever noticing a sensation, gently noting it, letting go, and continuing attending (5 minutes).
3. Being mindful of thought: Attending to mind, as thoughts come and go. Whenever a thought or feeling comes to mind, just noticing it, let go, and continuing attending, again and again and again (5 minutes).
4. Being mindful of sounds: Attending to the sounds one hears, without thinking about it. Just gently noticing it, letting it go, and continuing waiting (5 minutes).
5. Being mindful of taste. Imagining a wonderful bowl of pieces of favorite fruit and simply attending to a taste sensation, without thought, analysis, and effort (5 minutes)
6. Full meditation: Gently opening eyes and be mindful of the world of the moment. Quietly attending and waiting. When noticing something, be it a sight, sound, thought, or sensation, just letting it go and then resuming attending. Doing nothing. Waiting for what comes (5 minutes).

The experimental group received 30-minute of individually administered, guided, chairside intervention, during hemodialysis sessions. This protocol was found to be feasible, effective for patients on hemodialysis (Thomas, et al., 2017). Smith (2005) explained in his theory, called as the ABC relaxation theory, at least two and preferably five weekly 30-minute sessions of actual training of mind-body therapies should be provided to evoke relaxation, relieve stress, and improve health in general populations. However, for hemodialysis patients, it has been suggested that brief program formatting with at least 400 total minutes may lead greater health benefits for hemodialysis patients (Nassim, et al., 2021). Accordingly, the experimental group received 30 minutes of mindfulness meditation; 3 times a week for 5 weeks (450 minutes)

However, the participants received also 2-hour Foundation Course before actual training sessions by a study researcher, which taught the participants the basics, benefits, and protocol of intervention and the method of accessing the intervention. To ensure the consistent delivery of intervention, the researcher recorded the intervention instructions in Arabic language based on the Smith (2005) protocol and sent audio-recorded instructions to the participants by their WhatsApp application or emails. The audio-recorded intervention contents were validated by 2 psychologists and an expert in meditation. The recorded intervention instructions were used by the participants during sessions using their cell phone and headsets as recommended (Nassim, et al., 2021). This method allowed up to 3-5 participants to receive the instructions and perform the intervention simultaneously.

The researcher who was responsible for developing the study intervention and supervised the intervention delivery were an experienced mind-body practitioner who received a 4-day training of mindfulness meditation. The researcher attended the sessions to manage any potential interruption and evaluate the intervention delivery. The participants' privacy was maintained by using curtains surrounding each participant during intervention. The participants were asked not to share any information related to the intervention with the participants in the control group. Participants in the control group received treatment as usual in the hemodialysis setting.

3.6 Procedure

First, the study's instruments' consent to be utilized was sought. One of the study researchers (Albustanji A.) carried out the participant recruitment after receiving permission from the hospital officials to carry out the study. The patients were given a thorough explanation of the study's goals and protocol. Patients who completed the eligibility requirements and agreed to participate in the study were asked to sign a permission form. The baseline measurements were then completed by the participants, utilizing the self-report questionnaires (T0) for the study variables. To give the intervention to patients, a research assistant with a bachelor's in nursing, 15 years of nursing experience, a diploma in nephrology, and a master's in psychology was asked; however, she was not involved in the recruitment procedure, data collection, or randomization. Using a simple computer-generated sequence, randomly assigning the participants to the experimental group (n = 31) or the control group (n = 31). The research variables were assessed for both groups after two weeks of the intervention (T1) and at the finish of the last session (T2). The same research assistant, who was not involved in any other aspects of the study and was blinded to the randomized allocation, measured the study variables at T0, T1, and T2. Every measurement was done in privacy at the dialysis facility.

3.7 Data Analysis

Statistical analysis was conducted using SPSS software (version 23). Descriptive statistics were used to describe the sample. The sample and variables were described by measures of central tendency and dispersion appropriate to the level of measurement. For example, means and SD were calculated for the dependent variables that were measured on interval level of measurement, and frequency were calculated for the categorical variables such as gender. Initial analyses were conducted to ensure that the randomization across covariates was successful. The variables of gender, marital status, employment, renal failure length, and smoking, and comorbidities variables were all tested at baseline using Chi-square to demonstrate that they were not significantly different between groups.However, the variables of age and weight were tested at baseline using Independent t-tests to make sure the study groups were not significantly different on these variables before introducing mindfulness meditation.

Repeated measures(RM) ANOVA (within-subject only) were used to test the first study hypothesis. Repeated measures ANOVA for mixed designs (between-subjects and within-subjects designs) were used to test the second study hypothesis. The analysis compared means for the same people over time (within-subjects factor), means for different people in the treatment groups (between-subjects factor), as well as the interaction term (group X time factors). Post hoc t-tests were run to examine if the two study groups were significantly different on the dependent variables at the middle or end of the intervention separately.

3.8 Ethical Consideration

The Jordan University of Science and Technology institutional review board (IRB) and Ministry of health approved the procedure. After a full explanation of the study's purpose, procedures, benefits, and significance, the patient was asked to sign a consent form. Additionally, the subjects will be informed of their right to withdraw from the study at any time and the confidentiality and anonymity of their information. Each participant's anonymity will be maintained using a numeric code, and the study data will be stored. No patient was excluded from the study because of gender, ethnicity, or nationality. During the intervention, if the patient feels any complications, the intervention will be stopped.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patient receiving hemodialysis three times per week,
* being at least 18 years old,
* being able to read and write Arabic.

Exclusion Criteria:

* Patients with cognitive dysfunction or mental retardation,
* those who regularly used psychopharmacological, pain or sleeping pills,
* or received psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Pain perception | 6 weeks
  The Numeric Pain Rating Scale (NPRS) is a unidimensional measure of pain severity in adults (Child et al.,2005).The NPRS is a segmented numerical version of the visual analog scale (VAS), in which the respondent chooses a number (0-10 integers) that best describes the degree of pain (Rodriguez, 2001). Both literate and illiterate rheumatoid arthritis patients have shown high test-retest reliability (r = 0.96 and 0.95, respectively). For evaluating pain levels in Arabic countries, the Arabic Numeric Pain Rating Scale was a valid and reliable tool.The Arabic Numerical Pain Rating Scale had a high correlation coefficient (r140.93-0.94) with the VAS and VRS, indicating strong consistency in pain level measures among the three pain scales (Alghadir, Anwer, & Iqbal, 2016).
Quality of sleep | 6 weeks
  quality of sleep was measured by The Pittsburgh Sleep Quality Index (PSQI) (Buysse, Reynolds, Monk, Berman, and Kupfer, 1989). The PSQI was created to assess the clinical population's sleep quality. Subjective sleep quality (1 item), sleep latency (2 items), sleep duration (1 item), habitual sleep efficiency (3 items), sleep disturbances (9 items), use of sleeping medication (1 item), and daytime dysfunction (2) are the seven dimensions of sleep characteristics included in the PSQI. The scoring of PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty).
Self-esteem | 6 weeks
  self-esteem was measured by the Rosenberg self-esteem scale (Rosenberg, 1989). Total score range from 10-40, highest score reveals better self-esteem (Rosenberg, 1979). The Arabic version of the RSES is valid, reliable, and beneficial to use among the Arab community, according to two studies conducted among the Arab population in Jordan and Lebanon (Bezri et al., 2022).

CONTACTS AND LOCATIONS:
Overall Officials: Hossam Alhawatmeh, Principal Investigator — Hossam alhawatmeh, associate professor, Jordan university of science and technology
Locations (1):
- Jordan University of Science and Technology, Irbid, None Selected, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chu SWF, Yeam CT, Low LL, Tay WY, Foo WYM, Seng JJB. The role of mind-body interventions in pre-dialysis chronic kidney disease and dialysis patients - A systematic review of literature. Complement Ther Med. 2021 Mar;57:102652. doi: 10.1016/j.ctim.2020.102652. Epub 2020 Dec 26. PMID 33373760
- [Background] Shinde, M., & Mane, S. P. (2014). Stressors and the Coping Strategies among Patients Undergoing Hemodialysis, 3(2), 266-276.
- [Background] Jeong, M. H., & Park, O. L. (2012). Effects of dan jeon breathing on stress, sleep disturbance and self-esteem of Hemodialysis Patients. Journal of the korea academia-industrial cooperation society, 13(12), 5882-5892.
- [Background] Darvishi A, Otaghi M, Mami S. The Effectiveness of Spiritual Therapy on Spiritual Well-Being, Self-Esteem and Self-Efficacy in Patients on Hemodialysis. J Relig Health. 2020 Feb;59(1):277-288. doi: 10.1007/s10943-018-00750-1. PMID 30673996
- [Background] Alradaydeh, M. F., & Khalil, A. A. (2019). The effectiveness of physical exercise on psychological status, and sleep quality among jordanian patients undergoing hemodialysis: Literature review. Open Journal of Nursing, 9(12), 1267.
- [Background] Poorgholami F, Javadpour S, Saadatmand V, Jahromi MK. Effectiveness of Self-Care Education on the Enhancement of the Self-Esteem of Patients Undergoing Hemodialysis. Glob J Health Sci. 2015 Jun 12;8(2):132-6. doi: 10.5539/gjhs.v8n2p132. PMID 26383201
- [Background] Bennett PN, Ngo T, Kalife C, Schiller B. Improving wellbeing in patients undergoing dialysis: Can meditation help? Semin Dial. 2018 Jan;31(1):59-64. doi: 10.1111/sdi.12656. Epub 2017 Nov 2. PMID 29098724
- [Background] Rambod M, Sharif F, Pourali-Mohammadi N, Pasyar N, Rafii F. Evaluation of the effect of Benson's relaxation technique on pain and quality of life of haemodialysis patients: a randomized controlled trial. Int J Nurs Stud. 2014 Jul;51(7):964-73. doi: 10.1016/j.ijnurstu.2013.11.004. Epub 2013 Nov 25. PMID 24332569
- [Background] Al-Ghabeesh SH, Rayan A, Hattab F, Jarrar Y. Mindfulness and psychological distress among hemodialysis patients. Psychol Health Med. 2022 Apr;27(4):917-924. doi: 10.1080/13548506.2021.1960395. Epub 2021 Jul 28. PMID 34320891
- [Background] Rayan A, Ahmad M. The psychometric properties of the mindful attention awareness scale among Arab parents of children with autism spectrum disorder. Arch Psychiatr Nurs. 2018 Jun;32(3):444-448. doi: 10.1016/j.apnu.2018.01.001. Epub 2018 Jan 3. PMID 29784228
- [Background] Alhawatmeh H, Alshammari S, Rababah JA. Effects of mindfulness meditation on trait mindfulness, perceived stress, emotion regulation, and quality of life in hemodialysis patients: A randomized controlled trial. Int J Nurs Sci. 2022 Mar 8;9(2):139-146. doi: 10.1016/j.ijnss.2022.03.004. eCollection 2022 Apr. PMID 35509694
- [Background] Pai MF, Hsu SP, Yang SY, Ho TI, Lai CF, Peng YS. Sleep disturbance in chronic hemodialysis patients: the impact of depression and anemia. Ren Fail. 2007;29(6):673-7. doi: 10.1080/08860220701459642. PMID 17763161
- [Background] Dehghan M, Namjoo Z, Bahrami A, Tajedini H, Shamsaddini-Lori Z, Zarei A, Dehghani M, Ranjbar MS, Rafiee Sarbijan Nasab F. The use of complementary and alternative medicines, and quality of life in patients under hemodialysis: A survey in southeast Iran. Complement Ther Med. 2020 Jun;51:102431. doi: 10.1016/j.ctim.2020.102431. Epub 2020 May 21. PMID 32507442
- [Background] Razzera BN, Adamoli AN, Ranheiri MF, Oliveira MDS, Feoli AMP. Impacts of mindfulness-based interventions in people undergoing hemodialysis: a systematic review. J Bras Nefrol. 2022 Jan-Mar;44(1):84-96. doi: 10.1590/2175-8239-JBN-2021-0116. PMID 34643641
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777
- [Background] Alghadir AH, Anwer S, Iqbal ZA. The psychometric properties of an Arabic numeric pain rating scale for measuring osteoarthritis knee pain. Disabil Rehabil. 2016 Dec;38(24):2392-7. doi: 10.3109/09638288.2015.1129441. Epub 2016 Jan 6. PMID 26733318
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Rosenberg M, Court D. Regulatory sequences involved in the promotion and termination of RNA transcription. Annu Rev Genet. 1979;13:319-53. doi: 10.1146/annurev.ge.13.120179.001535. No abstract available. PMID 94251
- [Background] Nassim M, Park H, Dikaios E, Potes A, Elbaz S, Mc Veigh C, Lipman M, Novak M, Trinh E, Alam A, Suri RS, Thomas Z, Torres-Platas S, Vasudev A, Sasi N, Gautier M, Mucsi I, Noble H, Rej S. Brief Mindfulness Intervention vs. Health Enhancement Program for Patients Undergoing Dialysis: A Randomized Controlled Trial. Healthcare (Basel). 2021 Jun 1;9(6):659. doi: 10.3390/healthcare9060659. PMID 34205915
- [Background] Rodriguez-Amaya, D. B. (2001). A guide to carotenoid analysis in foods (Vol. 71). Washington: ILSI press.
- [Background] Bizri M, Kassir G, Tamim H, Kobeissy F, Hayek SE. Psychological distress experienced by physicians and nurses at a tertiary care center in Lebanon during the COVID-19 outbreak. J Health Psychol. 2022 May;27(6):1288-1300. doi: 10.1177/1359105321991630. Epub 2021 Feb 10. PMID 33567926